CLINICAL TRIAL: NCT04188769
Title: Effect of Local Pressure Application on Muscle Activity and General Relaxation in Persons With Hypertonia Following Stroke
Brief Title: Effect of Local Pressure on Muscle Activity and General Relaxation in Persons With Hypertonia Following Stroke
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of time
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EC/2019/1776
Record Dates: First submitted 2019-11-26; First posted 2019-12-06 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Deep Pressure; Muscle Activity; General Relaxation; Stroke; Hypertonia, Muscle
MeSH Terms: conditions — Stroke; Muscle Hypertonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- uninflated - rest (Sham Comparator): splint around the arm is not inflated both arms are in rest during the entire trial
  Interventions: Device: uninflated air splint
- uninflated - triggered (Sham Comparator): splint around the arm is not inflated 5x flexion and extension with the contralateral arm (with weight of 5kg in the hands)
  Interventions: Device: uninflated air splint; Other: contralateral movement
- constantly inflated - rest (Active Comparator): splint around the arm is constantly inflated both arms are in rest during the entire trial
  Interventions: Device: constant deep pressure applied by an air splint
- constantly inflated - triggered (Active Comparator): splint around the arm is constantly inflated 5x flexion and extension with the contralateral arm (with weight of 5kg in the hands)
  Interventions: Device: constant deep pressure applied by an air splint; Other: contralateral movement
- intermittently inflated - rest (Experimental): splint around the arm is intermittently inflated both arms are in rest during the entire trial
  Interventions: Device: intermittent deep pressure applied by an air splint
- intermittently inflated - triggered (Experimental): splint around the arm is intermittently inflated 5x flexion and extension with the contralateral arm (with weight of 5kg in the hands)
  Interventions: Device: intermittent deep pressure applied by an air splint; Other: contralateral movement

INTERVENTIONS:
Device: constant deep pressure applied by an air splint — inflation of the Johnstone air splint gives a constant local deep pression on the hemiplegic arm
  Arms: constantly inflated - rest; constantly inflated - triggered
Device: intermittent deep pressure applied by an air splint — continuous inflation and deflation of the Johnstone air splint gives an intermittent local deep pression on the hemiplegic arm
  Arms: intermittently inflated - rest; intermittently inflated - triggered
Device: uninflated air splint — no deep pressure applied by the air splint
  Arms: uninflated - rest; uninflated - triggered
Other: contralateral movement — non-hemiplegic arm is flexed and extended 5 times, with a weight of 5kg in the hand, in order to trigger hypertonia in the hemiplegic arm
  Arms: constantly inflated - triggered; intermittently inflated - triggered; uninflated - triggered

SUMMARY:
The purpose of this study is to examine the effect of - both constant as intermittent - local application of deep pressure on muscle activity and general relaxation in persons with hypertonia following stroke.

DETAILED DESCRIPTION:
This study will be carried out in 20 persons with hypertonia following stroke. There will be one single test occasion, during which 6 test trials will be performed in random order. Deep pressure will be applied by means of a Johnstone air splint, that will be (1) not inflated, (2) inflated constantly, or (3) inflated intermittently. Each of these 3 inflation conditions will be performed twice, i.e. with and without a non-hemiplegic arm movement (triggering hypertonia at hemiplegic side).

ELIGIBILITY:
Inclusion Criteria:

* subacute stroke (<6 months)
* hypertonia (Modified Ashworth Scale score of ≥2 for arm flexors at the hemiplegic side)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
EMG of biceps brachii | through study completion, an average of 5 months
  electromyographic frequency analysis of biceps brachii muscle activity at the hemiplegic side
EMG of triceps brachii | through study completion, an average of 5 months
  electromyographic frequency analysis of triceps brachii muscle activity at the hemiplegic side
EMG of pectoralis major | through study completion, an average of 5 months
  electromyographic frequency analysis of pectoralis major muscle activity at the hemiplegic side
MyotonPRO measurement of pectoralis major muscle tone | through study completion, an average of 5 months
  MyotonPRO measurement of pectoralis major muscle tone
heart rate | through study completion, an average of 5 months
  heart rate measurement assessed with the Zehpyr bioharness
heart rate variability | through study completion, an average of 5 months
  heart rate variability assessed with the Zehpyr bioharness
respiratory rate | through study completion, an average of 5 months
  respiratory rate assessed with the Zehpyr bioharness
subjective rating of hypertonia | through study completion, an average of 5 months
  visual analogue scale rating of the intensity of hypertonia, in which the degree of hypertonia has to be situated between "0" (no hypertonia) and "10" (very severe hypertonia)

SECONDARY OUTCOMES:
MyotonPRO measurement of pectoralis major elasticity | through study completion, an average of 5 months
  MyotonPRO measurement of pectoralis major elasticity
MyotonPRO measurement of pectoralis major stiffness | through study completion, an average of 5 months
  MyotonPRO measurement of pectoralis major stiffness

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided